CLINICAL TRIAL: NCT07243171
Title: A Multicenter, Multiple-dose Escalation, Randomized, Double-blind, Placebo-controlled Phase Ib/IIa Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral Ecnoglutide Tablets in Chinese Participants With Overweight or Obesity
Brief Title: A Phase Ib/IIa Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral Ecnoglutide Tablets in Chinese Participants With Overweight or Obesity
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hangzhou Sciwind Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCW0503-1012
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-10

CONDITIONS: Overweight and/or Obesity; Weight Management
Keywords: ecnoglutide; glucagon-like peptide-1 (GLP-1); obesity; overweight; weight management
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- oral ecnoglutide dose 1 (Experimental): once daily
  Interventions: Drug: ecnoglutide tablets
- oral ecnoglutide dose 2 (Experimental): once daily
  Interventions: Drug: ecnoglutide tablets
- oral ecnoglutide dose 3 (Experimental): once weekly
  Interventions: Drug: ecnoglutide tablets
- oral ecnoglutide dose 4 (Experimental): once weekly
  Interventions: Drug: ecnoglutide tablets
- placebo dose 1 (Placebo Comparator): once daily
  Interventions: Drug: placebo with matching dosage
- placebo dose 2 (Placebo Comparator): once weekly
  Interventions: Drug: placebo with matching dosage

INTERVENTIONS:
Drug: ecnoglutide tablets — oral tablets
  Arms: oral ecnoglutide dose 1; oral ecnoglutide dose 2; oral ecnoglutide dose 3; oral ecnoglutide dose 4
Drug: placebo with matching dosage — oral tablets
  Arms: placebo dose 1; placebo dose 2

SUMMARY:
The aim of the study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of oral ecnoglutide tablets in Chinese participants with overweight or obesity

DETAILED DESCRIPTION:
In this study, eligible participants will be randomized to receive either oral ecnoglutide tablet or placebo once daily for up to 3 weeks (Cohort C1) or 4 weeks (Cohort C2), or once weekly for up to 24 weeks (Cohort C3 and C4), including a dose escalation period.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of informed consent, with BMI in the range of 24.0 to 35.0 kg/m2 (including the threshold), body weight >60.0 kg for male, and weight >50.0 kg for female;
2. Self-declaration of body weight change <5% within 3 months prior to informed consent ;

Exclusion Criteria:

1. Diagnosis of overweight or obesity due to endocrine disorders , such as Cushing's syndrome;
2. Diagnosis of other endocrine disorders with clinical significance, including but not limited to hyperthyroidism or hypothyroidism, thyroid nodules (imaging shows TI-RADS≥ class 3), thyroid cancer, or personal or family history of type 2 multiple endocrine tumor syndrome (MEN2), etc.
3. Diagnosis of cardiovascular or cerebrovascular diseases with clinical significance within 6 months prior to screening, including but not limited to acute stroke, acute coronary syndrome, heart failure, arrhythmia, etc.
4. Diagnosis of severe gastrointestinal diseases, including but not limited to inflammatory bowel disease, active ulcers, irritable bowel syndrome, celiac disease, dyspepsia, diabetic gastroparesis, diabetic diarrhea, clinical gastric emptying abnormalities (such as pyloric obstruction), etc.
5. History of major gastrointestinal surgery (except cholecystectomy or appendectomy), or metabolic surgery, or plan to undergo major surgery during the study period;
6. HbA1c ≥6.5% or fasting blood glucose ≥7.0 mmol/L, or OGTT 2-hour blood glucose ≥11.1 mmol/L, at screening;
7. Clinical laboratory test results with clinical significance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-08-03 (Estimated); Study Completion 2026-11-22 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events | up to day 204

SECONDARY OUTCOMES:
Pharmacokinetics of oral ecnoglutide tablet | up to day 204
  Cmax, Tmax and AUC
Change of body weight from baseline | up to day 204
Change of BMI from baseline | up to day 204
Change of waist circumference from baseline | up to day 204
Change of hip circumference from baseline | up to day 204
Change of neck circumference from baseline | up to day 204
Change of waist/hip ratio from baseline | up to day 204
Change of fasting blood glucose from baseline | up to day 204
Change of fasting insulin from baseline | up to day 204
Change of lipid profile from baseline | up to day 204

OTHER OUTCOMES:
Immunogenecity of oral ecnoglutide tablet | up to day 204

CONTACTS AND LOCATIONS:
Overall Officials: Jintong Li, Dr, Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No